CLINICAL TRIAL: NCT04187300
Title: A Trial to Demonstrate Bioequivalence Between Semaglutide Formulation D With the DV3396 Pen-injector and Formulation B With the PDS290 Pen-injector in Subjects With Overweight or Obesity
Brief Title: A Research Study Looking at the Comparability (Bioequivalence) of Two Forms of Semaglutide in Two Different Pen-injectors in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9536-4590; U1111-1236-7697 (Other: World Health Organization (WHO)); 2019-002909-21 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV3396 (Experimental): Semaglutide administered with the DV3396 pen-injector (Formulation D)
  Interventions: Drug: Semaglutide
- PDS290 (Experimental): Semaglutide administered with the PDS290 pen-injector (Formulation B)
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Increasing doses of semaglutide administered s.c. (subcutaneouly, under the skin) once weekly for 20 weeks

SUMMARY:
The study will look at how two different forms of semaglutide reach and stay in the blood after injection. None of the two forms of semaglutide have been approved by the authorities to treat obesity, but it has been approved as a treatment for diabetes mellitus. Participants will get 1 of the 2 forms of semaglutide - which one is decided by chance. Participants will get the medicine as an injection under the skin of the belly using a pen-injector. The type of pen-injector is different for the two forms of semaglutide. The study staff will teach participants how to inject the medicine. Participants will take an injection once a week and will get a total of 21 injections of study medication. The study will last for about 27-30 weeks. Participants will have 25 study visits with the study doctor. For 2 of the visits, participants will stay in the clinic for 3 days and 2 nights. Participants may have to stop the study if the study doctor thinks that there are risks for their health. Women cannot take part if they are pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 27.0 and 34.9 kg/m^2 (both inclusive)
* Body weight between 70.0 and 130.0 kg (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Inability or unwillingness to perform self-injection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
AUC0-168h,2.4mg,SS, Area under the semaglutide concentration time curve | 0-168 hours (Day 141-148) after last 2.4 mg dose
  h*nmol/L
Cmax,2.4mg,SS, Maximum observed semaglutide concentration | 0-168 hours (Day 141-148) after last 2.4 mg dose
  nmol/L

SECONDARY OUTCOMES:
AUC0-168h,1mg,SS, Area under the semaglutide concentration time curve | 0-168 hours (Day 78-85) after last 1 mg dose
  h*nmol/L
Cmax,1mg,SS, Maximum observed semaglutide concentration | 0-168 hours (Day 78-85) after last 1 mg dose
  nmol/L
Tmax,2.4mg,SS, Time of maximum observed semaglutide concentration after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  h
Tmax,1mg,SS, Time of maximum observed semaglutide concentration after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  h
t½, terminal elimination half-life of semaglutide after last 2.4 mg dose | 0-1176 hours (Day 141-190) after last 2.4 mg dose
  h
Cl/F2.4mg, Total apparent clearance of semaglutide after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  L/h
Cl/F1mg, Total apparent clearance of semaglutide after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  L/h
Vss/F2.4mg, Apparent volume of distribution at steady-state of semaglutide after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  L
Vss/F1mg, Apparent volume of distribution at steady-state of semaglutide after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  L
Change in body weight | From baseline (Day 1, pre-dose) until the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com